CLINICAL TRIAL: NCT00492232
Title: Randomized, Double Blind, Placebo-Controlled Study to Assess Whether the Administration of Ramelteon Could Facilitate the Discontinuation of Zolpidem (Ambien®) ≥10 mg Therapy in Subjects With Chronic Insomnia
Brief Title: Facilitation of Zolpidem (≥10 mg) Discontinuation Through Use of Ramelteon in Subjects With Chronic Insomnia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-06-TL-375-071; U1111-1114-3262 (Registry Identifier: WHO)
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Results first posted 2009-07-17 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Chronic Insomnia
Keywords: Chronic Insomnia; Sleep Initiation and Maintenance Disorder; Drug Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — ramelteon; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramelteon 8 mg QD and current Zolpidem therapy (Experimental): Zolpidem therapy will be reduced by dose, frequency, or both for up to 10 weeks.
  Interventions: Drug: Ramelteon and zolpidem
- Placebo QD and current Zolpidem therapy (Placebo Comparator): Zolpidem therapy will be reduced by dose, frequency, or both for up to 10 weeks.
  Interventions: Drug: Placebo and zolpidem

INTERVENTIONS:
Drug: Ramelteon and zolpidem — Ramelteon 8 mg, tablets, orally, once daily and current zolpidem therapy incrementally reduced by dose, frequency, or both for up to 10 weeks.
  Other Names: Rozerem™; TAK-375; Ambien®
  Arms: Ramelteon 8 mg QD and current Zolpidem therapy
Drug: Placebo and zolpidem — Ramelteon placebo-matching tablets, orally, once daily and current zolpidem therapy incrementally reduced by dose, frequency, or both for up to 10 weeks.
  Other Names: Ambien®
  Arms: Placebo QD and current Zolpidem therapy

SUMMARY:
The purpose of this study is to assess whether ramelteon, once daily (QD), can facilitate the discontinuation of zolpidem in subjects with chronic insomnia.

DETAILED DESCRIPTION:
Approximately 60 to 70 million adults in the United States alone are affected by insomnia. Daytime symptoms of insomnia include tiredness, lack of energy, difficulty concentrating, and irritability. Recent epidemiologic research focusing on the quality of life has identified significant insomnia-related morbidities that relate to work productivity, health care utilization, and risk of depression. Insomnia is associated with diminished work output, absenteeism, and greater rates of accidents.

Zolpidem is the most commonly prescribed hypnotic in the United States for patients suffering from insomnia.

The purpose of this study is to assess whether ramelteon therapy can facilitate the discontinuation of benzodiazepine therapy in long term users. Subject participation in this study is anticipated to be about 17 weeks.

Subjects were screened and enrolled in a 4-week placebo run-in period, may have been randomized to a 10-week double-blind treatment period, and may have completed with a 2-week open-label treatment period. In the double-blind treatment period, subjects were randomized to one of two treatments: either ramelteon 8 mg tablets taken orally once-daily with concomitant current zolpidem therapy or to placebo-matching tablets once daily with concomitant current zolpidem therapy. Subjects incrementally reduced zolpidem therapy by dose, frequency, or both for up to 10 weeks. Only those subjects who completed the double-blind treatment period and had achieved a 50% reduction in zolpidem therapy during the double-blind treatment period participated in the open-label treatment period in which 8 mg ramelteon was administered. Zolpidem consumed during the open-label treatment period was recorded.

ELIGIBILITY:
Inclusion Criteria

* Chronic insomnia and taking greater than or equal to 10 mg zolpidem at least 4 times per week.
* Has been prescribed zolpidem for difficulty in initiating sleep.
* Must report chronic use of zolpidem greater than or equal to10 mg therapy for a minimum of 3 months prior to entry into Period 1 of the study.
* Must have taken zolpidem greater than or equal to 10 mg therapy for at least 4 of 7 days each week of the 4 weeks immediately prior to entry into the double blind phase, Period 2.
* Expressed a willingness to discontinue zolpidem therapy.
* Habitual bedtime is between 9:00 PM and 1:00 AM based on sleep history.
* Negative test result for hepatitis B surface antigen and hepatitis C virus antibody.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.

Exclusion Criteria

* Known hypersensitivity to ramelteon, zolpidem, or melatonin.
* Participated in any other investigational study and/or taken any investigational drug within 30 days prior to the first dose of run-in study medication.
* Sleep schedule changes required by employment (eg, shift worker) within 3 months prior to the first night of run-in study medication.
* History of fibromyalgia, history of seizures, sleep apnea, restless leg syndrome, periodic leg syndrome, chronic obstructive pulmonary disease, schizophrenia, bipolar disorder, mental retardation, or cognitive disorder.
* History of drug addiction or drug abuse within the past 12 months.
* History of alcohol abuse within the past 12 months, as defined in Diagnostic and Statistical Manual of Mental Disorders, 4th Edition revised and/or regularly consumes more than 2 alcoholic drinks per day.
* Current significant hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematological, or metabolic disease, unless currently controlled and stable with protocol-allowed medication, within 30 days prior to the first night of run-in study medication.
* Body mass index of less than 18 or greater than 34 (weight /height2).
* Any clinically important abnormal finding as documented by a medical history, physical examination, electrocardiogram, or clinical laboratory tests, as determined by the investigator.
* Positive hepatitis panel.
* Known history of human immunodeficiency virus.
* Any additional conditions(s) that in the investigator's opinion would affect:

  * sleep/wake function
  * prohibit the subject from completing the study
  * indicate that continuation in the study would not be in the best interests of the subject.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication, including:

  * Melatonin
  * Anxiolytics
  * Antipsychotics
  * Over-the-counter and prescription sedatives
  * Hypnotics (excluding zolpidem)
  * Narcotic analgesics
  * Antidepressants
  * Beta-blockers (exception is that Atenolol is permissible)
  * Anticonvulsants
  * St. John's wort
  * Sedating H1 antihistamines
  * Kava-kava
  * Systemic steroids
  * Ginkgo-biloba
  * Respiratory stimulants
  * Over-the-counter and prescription diet aids
  * Sedating Decongestants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2007-04; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda Global Research & Development Center
Locations (41):
- United States (41):
  - Hot Springs, Arkansas
  - Anaheim, California
  - Fountain Valley, California
  - La Mesa, California
  - Los Angeles, California
  - Redlands, California
  - San Diego, California
  - San Francisco, California
  - Santa Monica, California
  - Denver, Colorado
  - Clearwater, Florida
  - Hollywood, Florida
  - Kissimmee, Florida
  - Naples, Florida
  - Pembroke Pines, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Austell, Georgia
  - Boise, Idaho
  - Louisville, Kentucky
  - Metairie, Louisiana
  - Chevy Chase, Maryland
  - St Louis, Missouri
  - Lincoln, Nebraska
  - New York, New York
  - West Seneca, New York
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Greer, South Carolina
  - Fayetteville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Angelo, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah

REFERENCES:
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 38 investigative sites in the United States from 26 April 2007 to 28 May 2008.
Pre-assignment Details: Subjects completed a 4-week single-blind placebo run-in period prior to randomization in the double-blind treatment period (DBTP). During this time they took placebo-matching tablets once-daily (QD) with concomitant current zolpidem therapy. Subjects used a daily subject diary to record zolpidem dose reduction, daily activities, and sleep quality.
Groups:
- Ramelteon 8 mg QD: Ramelteon 8 mg, tablets, orally, once daily for up to 10 weeks in the DBTP.
- Placebo QD: Ramelteon placebo-matching tablets, orally, once daily for up to 10 weeks in the DBTP.
Period: Placebo Run-in
Arm/Group | Ramelteon 8 mg QD | Placebo QD
Started | 0 | 205 (All subjects received placebo in the placebo run-in period.)
Completed | 0 | 135 (These subjects successfully completed the placebo run-in period and were randomized to the DBTP.)
Not Completed | 0 | 70
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 0 | 3
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 0 | 8
Not completed — Pregnancy | 0 | 1
Not completed — Entrance criteria not met | 0 | 45
Not completed — Other | 0 | 6
Not completed — Missing | 0 | 2
Period: Double-Blind Treatment
Arm/Group | Ramelteon 8 mg QD | Placebo QD
Started | 65 | 70
Completed | 47 | 45
Not Completed | 18 | 25
Not completed — Adverse Event | 1 | 2
Not completed — Protocol Violation | 3 | 7
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 4 | 8
Not completed — Lack of Efficacy | 1 | 0
Not completed — Other | 6 | 5
Not completed — Randomized not treated | 1 | 0
Period: Open-Label Treatment
Arm/Group | Ramelteon 8 mg QD | Placebo QD
Started | 89 (In the previous DBTP, 45 and 44 subjects were randomized to ramelteon and placebo, respectively.) | 0 (All subjects received ramelteon in the OLTP.)
Completed | 88 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramelteon 8 mg QD | Placebo QD | Total
Number analyzed (Participants) | 65 | 70 | 135
Age Continuous [Mean (Standard Deviation); unit: years] | 51.5 (13.45) | 47.0 (12.98) | 49.2 (13.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 49 | 91.0
  Male | 23 | 21 | 44.0
Race/Ethnicity, Customized [Number; unit: Subjects]
  Asian | 1 | 1 | 2.0
  Black or African American | 5 | 9 | 14.0
  White | 59 | 59 | 118.0
  Multiracial | 0 | 1 | 1.0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 19.0
  Not Hispanic or Latino | 55 | 61 | 116.0
  Unknown or Not Reported | 0 | 0 | 0.0
Baseline average total daily zolpidem dosage [Number; unit: subjects]
  ≤10 mg | 56 | 60 | 116
  >10 mg | 8 | 10 | 18
  Information not available | 1 | 0 | 1
Use of pharmacological assistance to sleep [Number; unit: subjects] — Randomized subjects responded to the question, "How often per week do you use pharmacological assistance to sleep?" 4=4 nights/week; >4=5-7 nights/week.
  subjects
    4 nights per week | 8 | 9 | 17
    >4 nights per week | 57 | 61 | 118
Weekly frequency zolpidem consumption [Number; unit: subjects] — The average number of nights per week subjects took zolpidem was calculated.
  subjects
    0-3 nights per week | 0 | 0 | 0
    4 nights per week | 2 | 1 | 3
    5 nights per week | 8 | 9 | 17
    6 nights per week | 8 | 7 | 15
    7 nights per week | 46 | 53 | 99
    Information not available | 1 | 0 | 1
Baseline weekly zolpidem dosage [Mean (Standard Deviation); unit: Dosage (mg)] — Baseline for the weekly zolpidem dosage was calculated as the total amount zolpidem intake recorded by a subject during placebo run-in, divided by the number of days in the period, multiplied by 7. Ramelteon 8 mg n=64; Placebo n=70.
  Dosage (mg) | 68.7 (17.71) | 70.3 (20.37) | 69.5 (19.09)
Weekly frequency zolpidem consumption [Mean (Standard Deviation); unit: nights per week] — Average number of nights per week randomized subjects used zolpidem. Ramelteon 8 mg n=64; Placebo n=70.
  nights per week | 6.53 (0.835) | 6.60 (0.769) | 6.57 (0.799)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Discontinued Zolpidem Therapy
Description: Participants reduced zolpidem incrementally from Week 3 to Week 10 of the double-blind treatment period (DBTP). A participant who did not take any zolpidem during the last 7 days of the DBTP was defined as having completely discontinued zolpidem by that time point. The number of subjects who discontinued zolpidem at the end of the DBTP was summarized.
Time Frame: Week 10
Population: Analysis was performed on all randomized subjects who took at least 1 dose of study drug, who had completed the DBTP, and who had sufficient zolpidem dosage data in the last 7 days of the DBTP.
Measure: Number; unit: Percentage of participants
Arm/Group | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 52 | 49
Percentage of participants | 28.8 | 32.7
Statistical Analysis 1: Comparison: Ramelteon 8 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.484, Regression, Logistic — Statistical significance was determined at the 0.05 level; Log odds of achieving response were estimated using the logistic regression analysis adjusted for effects of treatment and pooled center; Adjusted Odds Ratio = 0.71, 95% CI [0.27 to 1.85]

2. Secondary Outcome: Change From Baseline in Weekly Zolpidem Dosage During Weeks 1-2
Description: Dosages of zolpidem taken were recorded during Weeks 1-2 of the DBTP. Differences in dosages from baseline were summarized. Weekly dosage was calculated as total amount of zolpidem taken divided by the number of days within the phase, multiplied by 7.
Time Frame: Baseline and Weeks 1-2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Dose (mg)
Arm/Group | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 52 | 49
Dose (mg) | -11.8 (3.06) | -11.6 (3.11)
Statistical Analysis 1: Comparison: Ramelteon 8 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.946, ANCOVA — P-values are from t-tests of the analysis of covariance (ANCOVA) model for the difference in least squares (LS) means between treatments. Statistical significance was determined at the 0.05 level; LS means are from an ANCOVA model with baseline zolpidem dosage (≤10 mg vs >10 mg) and pooled center as covariates; Mean Difference (Final Values) = -0.2, 95% CI [-6.23 to 5.81]

3. Secondary Outcome: Change From Baseline in Weekly Zolpidem Dosage During Weeks 3-4
Description: Dosages of zolpidem taken were recorded during Weeks 3-4 of the DBTP. Differences in dosages from baseline were summarized. Weekly dosage was calculated as total amount of zolpidem taken divided by the number of days within the phase, multiplied by 7.
Time Frame: Baseline and Weeks 3-4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Dose (mg)
Arm/Group | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 52 | 49
Dose (mg) | -35.3 (2.89) | -35.6 (2.93)
Statistical Analysis 1: Comparison: Ramelteon 8 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.901, ANCOVA — P-values are from t-tests of the ANCOVA model for the difference in LS means between treatments. Statistical significance was determined at the 0.05 level; LS means are from an ANCOVA model with baseline zolpidem dosage (≤10 mg vs >10 mg) and pooled center as covariates; Mean Difference (Final Values) = 0.4, 95% CI [-5.31 to 6.03]

4. Secondary Outcome: Change From Baseline in Weekly Zolpidem Dosage During Weeks 5-6
Description: Dosages of zolpidem taken were recorded during Weeks 5-6 of the DBTP. Differences in dosages from baseline were summarized. Weekly dosage was calculated as total amount of zolpidem taken divided by the number of days within the phase, multiplied by 7.
Time Frame: Baseline and Weeks 5-6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Dose (mg)
Arm/Group | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 52 | 48
Dose (mg) | -40.2 (3.18) | -42.1 (3.22)
Statistical Analysis 1: Comparison: Ramelteon 8 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.538, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS means are from an ANCOVA model with baseline zolpidem dosage (≤10 mg vs >10 mg) and pooled center as covariates; Mean Difference (Final Values) = 2.0, 95% CI [-4.32 to 8.23]

5. Secondary Outcome: Change From Baseline in Weekly Zolpidem Dosage During Weeks 7-8
Description: Dosages of zolpidem taken were recorded during Weeks 7-8 of the double blind period. Differences in dosages from baseline were summarized.
Time Frame: Baseline and Weeks 7-8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Dose (mg)
Arm/Group | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 51 | 48
Dose (mg) | -52.1 (3.49) | -49.9 (3.49)
Statistical Analysis 1: Comparison: Ramelteon 8 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.517, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS means are from an ANCOVA model with baseline zolpidem dosage (≤10 mg vs >10 mg) and pooled center as covariates; Mean Difference (Final Values) = -2.2, 95% CI [-9.09 to 4.60]

6. Secondary Outcome: Change From Baseline in Weekly Zolpidem Dosage During Weeks 9-10
Description: Dosages of zolpidem taken were recorded during Weeks 9-10 of the DBTP. Differences in dosages from baseline were summarized. Weekly dosage was calculated as total amount of zolpidem taken divided by the number of days within the phase, multiplied by 7.
Time Frame: Baseline and Weeks 9-10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Dose (mg)
Arm/Group | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 52 | 49
Dose (mg) | -60.6 (3.27) | -60.7 (3.31)
Statistical Analysis 1: Comparison: Ramelteon 8 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.965, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS means are from an ANCOVA model with baseline zolpidem dosage (≤10 mg vs >10 mg) and pooled center as covariates; Mean Difference (Final Values) = 0.1, 95% CI [-6.28 to 6.56]

7. Secondary Outcome: Change From Baseline in Weekly Zolpidem Frequency During Weeks 1-2
Description: The number of nights zolpidem was taken was recorded during Weeks 1-2 of the DBTP. Weekly frequency was calculated as the number of nights zolpidem was taken divided by the number of days within the period, multiplied by 7. Differences in frequency from BL were summarized.
Time Frame: Baseline and Weeks 1-2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nights per week
Arm/Group | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 52 | 49
nights per week | 0.13 (0.183) | 0.04 (0.186)
Statistical Analysis 1: Comparison: Ramelteon 8 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.617, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS means are from an ANCOVA model with baseline zolpidem dosage (≤10 mg vs >10 mg), baseline zolpidem frequency, and pooled center as covariates; Mean Difference (Final Values) = 0.09, 95% CI [-0.27 to 0.45]

8. Secondary Outcome: Change From Baseline in Weekly Zolpidem Frequency During Weeks 3-4
Description: The number of nights zolpidem was taken was recorded during Weeks 3-4 of the DBTP. Weekly frequency was calculated as the number of nights zolpidem was taken divided by the number of days within the period, multiplied by 7. Differences in frequency from baseline were summarized.
Time Frame: Weeks 3-4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nights per week
Arm/Group | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 52 | 49
nights per week | -0.08 (0.288) | -0.26 (0.292)
Statistical Analysis 1: Comparison: Ramelteon 8 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.541, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 0.17, 95% CI [-0.39 to 0.74]

9. Secondary Outcome: Change From Baseline in Weekly Zolpidem Frequency During Weeks 5-6
Description: The number of nights zolpidem was taken was recorded during Weeks 5-6 of the DBTP. Weekly frequency was calculated as the number of nights zolpidem was taken divided by the number of days within the period, multiplied by 7. Differences in frequency from baseline were summarized.
Time Frame: Weeks 5-6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nights per week
Arm/Group | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 52 | 48
nights per week | -0.05 (0.396) | -0.60 (0.400)
Statistical Analysis 1: Comparison: Ramelteon 8 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.163, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 0.55, 95% CI [-0.23 to 1.33]

10. Secondary Outcome: Change From Baseline in Weekly Zolpidem Frequency During Weeks 7-8
Description: The number of nights zolpidem was taken was recorded during Weeks 7-8 of the DBTP. Weekly frequency was calculated as the number of nights zolpidem was taken divided by the number of days within the period, multiplied by 7. Differences in frequency from baseline were summarized.
Time Frame: Baseline and Weeks 7-8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nights per week
Arm/Group | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 51 | 48
nights per week | -1.10 (0.475) | -1.24 (0.475)
Statistical Analysis 1: Comparison: Ramelteon 8 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.757, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 0.15, 95% CI [-0.79 to 1.08]

11. Secondary Outcome: Change From Baseline in Weekly Zolpidem Frequency During Weeks 9-10
Description: The number of nights zolpidem was taken was recorded during Weeks 9-10 of the DBTP. Weekly frequency was calculated as the number of nights zolpidem was taken divided by the number of days within the period, multiplied by 7. Differences in frequency from baseline were summarized.
Time Frame: Baseline and Weeks 9-10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nights per week
Arm/Group | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 52 | 49
nights per week | -2.22 (0.534) | -2.34 (0.542)
Statistical Analysis 1: Comparison: Ramelteon 8 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.820, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 0.12, 95% CI [-0.93 to 1.17]

12. Secondary Outcome: Participants Who Completely Discontinued Zolpidem at the End of Double-Blind Treatment Period, by Method of Discontinuation
Description: Participants who took no zolpidem during the last 7 days of the DBTP were completely discontinued from zolpidem. Participants who completely discontinued zolpidem via reduction in zolpidem use frequency (alone) were not summarized.
Time Frame: Weeks 1-10
Population: Analysis was performed on all randomized subjects who took at least 1 dose of study drug, had completed the DBTP, and had sufficient zolpidem dosage data in the last 7 days of the DBTP. Estimates could not be reported with correct statistical inference due to small sample sizes by method of discontinuation (ie, most subjects reduced zolpidem dose).
Measure: Number; unit: participants
Arm/Group | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 52 | 49
participants
  Reduction in Dose | 12 | 8
  Reduction in Dose and Frequency | 3 | 8

13. Secondary Outcome: Participants Who Achieved a 50% Reduction in Zolpidem Dosage at the End of the Double-Blind Treatment Period
Description: Participants who achieved a 50% reduction in zolpidem dosage (or frequency) at the end of the DBTP (ie, the end of Reduction Phase 4) were summarized. The reduction in dosage at Reduction Phase 4=[1-(Reduction Phase 4 weekly dosage/baseline weekly dosage)]*100%.
Time Frame: Baseline and Week 10
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 52 | 49
participants | 48 | 42
Statistical Analysis 1: Comparison: Ramelteon 8 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.284, Regression, Logistic — P-values are from Chi-square tests of the log-regression model for the overall treatment comparison. Statistical significance was determined at the 0.05 level; Log odds of achieving response were estimated using logistic regression analysis adjusted for effects of baseline zolpidem dosage (≤10 mg vs >10 mg); Adjusted Odds Ratio = 2.01, 95% CI [0.55 to 7.34]

14. Secondary Outcome: Participants Who Achieved a 50% Reduction in Zolpidem Dosage at Any Time During the Double-Blind Treatment Period
Description: Participants who achieved a 50% reduction in zolpidem dosage at any previously defined 2-week period (ie, reduction phase) during the DBTP were summarized. The reduction in dosage at any time=[1-(reduction phase weekly dosage/baseline weekly dosage)]*100%.
Time Frame: Baseline and Weeks 1-10
Population: Analysis was performed on all subjects who were randomized and received at least 1 dose of double-blind medication during the study. Subjects were analyzed by the treatment they were randomized to receive.
Measure: Number; unit: participants
Arm/Group | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 64 | 70
participants | 50 | 50
Statistical Analysis 1: Comparison: Ramelteon 8 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.389, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; [statistical method as in outcome 13, analysis 1]; Adjusted Odds Ratio = 1.42, 95% CI [0.64 to 3.13]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events with onset dates the same or after the start of double-blind study medication and before the first dose of open-label study medication were summarized for the double-blind medication.
Description: Two ramelteon-treated subjects permanently discontinued the study due to adverse events during the double-blind treatment period. One placebo-treated subject had multiple temporary study drug interruptions due to adverse events but did not permanently discontinue the study
Arm/Group | Ramelteon 8 mg QD | Placebo QD
Serious Adverse Events (participants affected / at risk) | 0/64 | 1/70
Other Adverse Events (participants affected / at risk) | 11/64 | 7/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramelteon 8 mg QD (N=64) | Placebo QD (N=70)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramelteon 8 mg QD (N=64) | Placebo QD (N=70)
Upper Respiratory Tract Infections (Infections and infestations) | 5 (5) | 2 (2)
Dizziness (Nervous system disorders) | 4 (5) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period up to 150 days to permit actions necessary to preserve sponsor's intellectual property; can request changes to the results communication only for the purpose of removing non study related information that is proprietary and confidential to sponsor; can require delay of a results communication until the study has been completed at all participating sites.